CLINICAL TRIAL: NCT00006014
Title: A Phase II Trial of SU5416 (NSC# 696819) in Patients With Malignant Mesothelioma
Brief Title: SU5416 in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02351; UCCRC-10409; UCCRC-NCI-44; NCI-44; CDR0000068023 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2004-02-26 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2009-02

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma; epithelial mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Semaxinib

ARMS (1):
- Arm I (Experimental): Patients receive SU5416 IV over 1 hour twice weekly. Courses repeat every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: semaxanib

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
Phase II trial to study the effectiveness of SU5416 in treating patients who have malignant mesothelioma. SU5416 may stop the growth of malignant mesothelioma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate, median and overall survival, and time to progression in patients with unresectable malignant mesothelioma treated with SU5416.

II. Determine the effect of SU5416 on surrogate biologic endpoints, including microvessel density, tissue proliferative index, apoptosis, vascular endothelial growth factor levels, and tumor perfusion measured by MRI in these patients.

III. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive SU5416 IV over 1 hour twice weekly. Courses repeat every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 21-45 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven malignant mesothelioma (epithelial, sarcomatoid, or mixed subtype) that is not amenable to surgery or radiotherapy
* Measurable disease
* At least 20 mm by conventional techniques or at least 10 mm by spiral CT scan
* Pleural effusions and ascites are not considered measurable lesions
* Only site of measurable disease must not be located within prior radiotherapy port
* Lesion must be accessible for biopsy
* History of previously treated CNS metastasis allowed if:

  * Neurologically stable
  * No requirement for IV or oral steroids or IV anticonvulsants
  * No active or residual disease by brain CT or MRI scan
* Patients with neurologic signs or symptoms suggestive of CNS metastasis must have a negative brain CT or MRI scan

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: WHO 0-2
* Life expectancy: At least 12 weeks
* WBC at least 3,000/mm3
* Platelet count at least 75,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* No uncompensated coronary artery disease on electrocardiogram or physical examination
* No history of myocardial infarction or severe/unstable angina within the past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No deep vein or arterial thrombosis within the past 3 months
* No pulmonary embolism within the past 3 months
* No significant uncontrolled underlying medical or psychiatric illness
* No serious active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active second malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Patients are not considered to have active malignancy if they have completed therapy and are considered to be at less than 30% risk of relapse
* No history of severe allergic or anaphylactic reactions to paclitaxel or docetaxel

PRIOR CONCURRENT THERAPY:

* No more than 1 prior systemic chemotherapy regimen
* At least 4 weeks since prior systemic chemotherapy and recovered
* Prior intrapleural cytotoxic agents (including bleomycin) allowed
* No concurrent chemotherapy
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* At least 30 days since prior investigational drug and recovered
* No concurrent investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2000-08; Primary Completion 2007-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana